CLINICAL TRIAL: NCT05544825
Title: Evaluation of Efficacy and Safety of Ice Plant (Mesembryanthemum Crystallinum) Extract in Patients With Impaired Fasting Glucose: a Double-blind, Randomized, Placebo-controlled Study
Brief Title: Ice Plant (Mesembryanthemum Crystallinum) Extract in Patients With Impaired Fasting Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2022-016
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Impaired Fasting Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ice plant group (Experimental): This group takes ice plant extract for 12 weeks.
  Interventions: Dietary Supplement: Ice plant group
- Placebo group (Placebo Comparator): This group takes a placebo for 12 weeks.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Ice plant group — Ice plant extract 2,000 mg/day for 12 weeks
  Arms: Ice plant group
Dietary Supplement: Placebo group — Placebo 2,000 mg/day for 12 weeks
  Arms: Placebo group

SUMMARY:
The investigators will conduct a randomized, double-blind, placebo-controlled study to investigate the effects and tolerability of ice plant (Mesembryanthemum crystallinum) extract in patients with impaired fasting glucose for 12 weeks.

DETAILED DESCRIPTION:
A previous animal study has indicated that ice plant (Mesembryanthemum crystallinum) extract (IPE) has a substantial effect on attenuating hyperglycemia and modulating gut microbiota composition in diabetic rats. Therefore, IPE might be a promising functional food for the prevention of diabetes. Therefore, the investigators will conduct a randomized, double-blind, placebo-controlled study to investigate the effects of IPE in patients with impaired fasting glucose for 12 weeks; the safety of the compound is also evaluated. The Investigators examine 75-g oral glucose tolerance test (OGTT) (120 minute glucose), 75-g OGTT incremental Area Under the Curve 0-120min, 75-g OGTT (0, 30, 60, 90 minute glucose), fasting insulin, Homeostasis Model Assessment for Insulin Resistance, Quantitative Insulin Sensitivity Check Index, HbA1c, lipid profile (total cholesterol, triglyceride, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol) at baseline and after 12 weeks of intervention. One hundred adults were administered either 2,000 mg of IPE or a placebo each day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Those with fasting blood glucose of 100 mg/dL or more and less than 140 mg/dL

Exclusion Criteria:

* Those who have been diagnosed with type 1 or type 2 diabetes
* Those who have continuously taken drugs that may affect blood glucose, such as blood glucose-lowering drugs or anti-obesity drugs, within 3 months
* A person who has continuously taken health functional food that can affect blood glucose within 1 month or health functional food can affect the interpretation of the results of this study
* Those who took systemic steroids within 1 month
* Those who lost 0% or more in weight within the last 3 months
* Severe cerebrovascular disease (cerebral infarction, cerebral hemorrhage, etc.) within the last 6 months), heart disease (angina pectoris, myocardial infarction, heart failure, arrhythmia that needs to be treated), or a malignant tumor (however, subjects with a history of cerebrovascular disease or heart disease but clinically stable are not eligible for the study at the discretion of the investigator.
* Persons with local or systemic inflammatory diseases
* Persons with renal disease such as hereditary hyperlipidemia, acute/chronic renal failure, nephrotic syndrome
* Persons with systolic blood pressure (BP) 160mmHg or diastolic BP 100mmHg or higher (provided that, those who are stably controlling their BP through drug treatment can participate)
* Those with HbAc1 of 7.0% or higher
* Abnormal liver or renal function (more than twice the normal upper limit of the research institute)
* Those who are currently being treated for thyroid disease
* Those who have a history of gastrointestinal disease (eg, Crohn's disease) or gastrointestinal surgery (except simple appendectomy or hernia surgery) that may affect the absorption of the test food
* Those who have participated or plan to participate in other drug clinical trials within the last 1 month
* Persons taking drugs for psychiatric disorders (except for cases of intermittent medication due to sleep disturbance)
* Persons with alcoholism, drug abuse, or dependence
* Pregnant or lactating or during this human application test period Women who plan to become pregnant during pregnancy
* Those who have a clinically significant history or allergic reaction to drugs or food for human application
* Appropriate methods of contraception among women of childbearing age (condoms, diaphragms, intrauterine contraceptives, male partner Women who do not accept the procedure (if they have undergone resection) (however, women who have undergone sterilization are excluded)

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
75-g Oral Glucose Tolerance Test (120 minute glucose) | 12 weeks
  mg/dL

SECONDARY OUTCOMES:
Incremental Area Under the Curve 0-120 minutes | 12 weeks
  mg/dL
75-g Oral Glucose Tolerance Test (0, 30, 60, 90 minute glucose) | 12 weeks
  mg/dL
Fasting Insulin | 12 weeks
  µU/ml
Homeostasis Model Assessment for Insulin Resistance | 12 weeks
  fasting insulin (µU/ml) + fasting glucose (mg/dl)/405
Quantitative Insulin Sensitivity Check Index | 12 weeks
  1/(log(fasting insulin µU/ml) + log(fasting glucose mg/dl))
HbA1c | 12 weeks
  percentage
Total cholesterol | 12 weeks
  mg/dL
Triglyceride | 12 weeks
  mg/dL
Low-density lipoprotein cholesterol | 12 weeks
  mg/dL
High-density lipoprotein cholesterol | 12 weeks
  mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea